CLINICAL TRIAL: NCT05266677
Title: Effect of a Liquid Oral Supplement Comprising a Blend of Glycerides at Certain Proportions on Infant and Toddler DHA Status
Brief Title: DHA Proof-of-Concept Study in Infants and Toddlers
Acronym: DHA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Foreseen high level of subject burden and non compliance in the clinical trial due to extensive product preparation and the nutritional concept for the improvement of RBC DHA is compromised by the change in the product formulation
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 18.20.NRC
Record Dates: First submitted 2022-01-04; First posted 2022-03-04 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Infants; Toddlers; Nutritional Supplement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPL (Experimental): Liquid oral supplement comprising a blend of glycerides at certain proportions
  Interventions: Other: blend of glycerides at certain proportions
- CTRL (Other): Liquid oral supplement comprising glycerides used in current formulas
  Interventions: Other: glycerides used in current formulas

INTERVENTIONS:
Other: blend of glycerides at certain proportions — combination of glycerides in specific proportions in a liquid oral supplement
  Arms: EXPL
Other: glycerides used in current formulas — glycerides used in current formulas in a liquid oral supplement
  Arms: CTRL

SUMMARY:
This is a prospective, double blind, randomized, controlled proof-of-concept study with a parallel group design that aims to investigate the effect of a liquid oral supplement comprising a blend of glycerides at certain proportions on infant and toddler DHA status.

ELIGIBILITY:
Inclusion Criteria:

Subjects who fulfil all of the following inclusion criteria will be included:

1. Evidence of personally signed and dated informed consent form indicating that the infant/toddler's parent(s)/ Legally Authorized representative (LAR) has been informed of all pertinent aspects of the study.
2. Infants/toddlers whose parent(s)/LAR are willing and able to comply with scheduled visits, and the requirements of the study protocol.
3. Infants/toddlers must meet the following inclusion criteria respectively to be eligible for enrollment into the study:

   1. Healthy normally developing infant/toddler at the discretion of the investigator.
   2. Healthy term infant (37-42 weeks of gestation) at birth.
   3. At enrollment visit, post-natal age 2-3 months (60-90 days) for infants or 13-14 months for toddlers (date of birth = day 0).
   4. For the infant group, infants must have been exclusively consuming and tolerating a cow's milk infant formula not containing DHA for the past month, and their parent(s)/LAR must have independently elected, before enrolment, not to breastfeed.
   5. For the toddler group, toddlers must have been consuming and tolerating a cow's milk TMS not containing DHA for the past month.
   6. Infants or toddlers must not have been consuming DHA-containing supplements for the past month.

Exclusion Criteria:

Any of the following criteria would render a subject ineligible for inclusion:

1. Infants/toddlers with conditions requiring feedings other than those specified in the protocol.
2. Infants receiving complementary foods or liquids defined as 4 or more teaspoons per day or approximately 20 grams (g) per day of complementary foods or liquids at enrollment.
3. Infants/toddlers who have a medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results, including:

   1. Evidence of major congenital malformations (e.g., cleft palate, extremity malformation).
   2. Suspected or documented systemic or congenital infections (e.g., human immunodeficiency virus, cytomegalovirus, syphilis).
   3. Evidence of significant cardiac, respiratory, endocrinologic, hematologic, gastrointestinal (e.g., complicated gastroesophageal reflux combined with inadequate growth and/or respiratory complications, Hirschsprung's disease), or other systemic diseases.
   4. History of admission to the Neonatal Intensive Care Unit, with the exception of admission for jaundice phototherapy.
   5. Currently participating or having participated in another clinical trial since birth.
   6. Other severe medical or laboratory abnormality (acute or chronic) which, in the judgment of the investigator, would make the infant/toddler inappropriate for entry into the study.
4. Infants/toddlers who are presently receiving or have received prior to enrollment any of the following: medication(s) or supplement(s) which are known or suspected to affect fat digestion, absorption, and/or metabolism (e.g., lactase enzymes, pancreatic enzymes); medications that may neutralize or suppress gastric acid secretion; medications that could affect any study outcomes.
5. Infants/toddlers whose parent(s)/LAR who in the Investigator's assessment cannot be expected to comply with the protocol or with study procedures.

Ages: 2 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
RBC-DHA levels after 56 days of supplementation | Study day 56
  Red blood cell (RBC)-DHA after eight weeks of intervention

SECONDARY OUTCOMES:
RBC, plasma additional fatty acids status | Study days 0, 14, 28 and 56
  Determination of omega-3, omega-6, eicosapentanoic acid, arachidonic acid
DHA supplement intake | Study days 3, 14, 28 and 56
  Parent-reported supplement intake assessed using a 3-day DHA Supplement Intake and Tolerance Diary
Gastrointestinal (GI) tolerance | Study days 3, 14, 28 and 56
  Parent-reported GI tolerance indicators assessed using a 3-day DHA Supplement Intake and Tolerance Diary
Weight | Study days 0, 14, 28 and 56
  Weight measured in grams
Length | Study days 0, 14, 28 and 56
  Length measured in cm
Head circumference | Study days 0, 14, 28 and 56
  Head circumference measured in cm
Dietary intakes of DHA and other fatty acids (toddler population only) | Study days 0, 28 and 56
  Assessed using a 24-hour food recall
Standard adverse events (AEs) and serious AEs (SAEs) reporting for safety assessment | Study days 0, 14, 28, 56, and 70
  Incidence of AEs / SAEs reported throughout the study, particular attention will be paid to AEs related to GI tolerance and comfort

CONTACTS AND LOCATIONS:
Overall Officials: Elvira M Estorninos, MD, Principal Investigator — Las Pinas Doctors Hospital

IPD SHARING:
Plan to Share IPD: No